CLINICAL TRIAL: NCT05842980
Title: BIomarkers to Predict the Outcomes of Sepsis
Acronym: BIPROS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: BIPROS
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Sepsis
Keywords: sepsis; biomarker
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5ml blood from sepsis patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sepsis: sepsis patients
  Interventions: Other: sepsis

INTERVENTIONS:
Other: sepsis — collect 5ml blood from patient

SUMMARY:
Sepsis is an organ dysfunction syndrome caused by the host's immune response to infection, and is one of the common critical illnesses. However, sepsis remains the main threat to global health. Due to the high heterogeneity, the diagnosis of sepsis is difficult, and it is particularly important to find biomarkers that can predict changes in the patient's condition and prognosis. The purpose of this study is to collect patient blood samples for testing and identify biomarkers related to the prognosis of sepsis.

DETAILED DESCRIPTION:
Sepsis is an organ dysfunction syndrome caused by the host's immune response to infection, and is one of the common critical illnesses. There are reports that the mortality rate of sepsis patients is 25-30%, and the hospital mortality rate of septic shock is as high as 40-60%. According to Lancet data, in 2017, there were 48.9 million cases of sepsis worldwide, resulting in approximately 11 million deaths, accounting for 19.7% of the total global deaths. Surviving sepsis patients often experience secondary infections and chronic organ dysfunction, which affects their long-term quality of life and poses a huge socio-economic burden. The World Health Organization (WHO) has identified sepsis as a global health priority and called for improving the level of sepsis prevention and treatment. With the advancement of medical technology, the diagnostic and treatment guidelines for sepsis are constantly updated, and clinical treatment capabilities have been improved. However, sepsis remains the main threat to global health. Due to the high heterogeneity, the diagnosis of sepsis is difficult, and it is particularly important to find biomarkers that can predict changes in the patient's condition and prognosis. The purpose of this study is to collect patient blood samples for testing and identify biomarkers related to the prognosis of sepsis.

ELIGIBILITY:
Inclusion Criteria:

-

The clinical diagnostic criteria for sepsis or septic shock that comply with the 3rd edition of the International Consensus on Sepsis and Sepsis Shock (Sepsis-3.0) are:

1. Sepsis-3.0 sepsis diagnosis criteria: infection or suspected infection with a Sequential Organ Failure Score (SOFA score) ≥ 2 points;
2. Sepsis-3.0 diagnostic criteria for septic shock: Sepsis with persistent hypotension, after sufficient fluid resuscitation, still requires vasopressor drugs to maintain average arterial pressure ≥ 65mmHg, and serum lactate level>2mmol/L (18mg/dL).
3. Age 18 to 85 years old

Exclusion Criteria:

1. patients with autoimmune disease, acquired immunodeficiency syndrome, agranulocytosis (<0.5 × 109/L), malignant tumors or other serious chronic diseases (heart failure, Liver failure, end-stage renal disease, etc.);
2. Receiving glucocorticoid treatment;
3. Pregnancy;
4. Refuse enrollment or give up active treatment. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion of patients diagnosed with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
28d all-cause mortality | 28 days
  28d all-cause mortality

SECONDARY OUTCOMES:
Incidence of secondary infection | Day 0 to 28
  recurrence, double infection and new infection
ICU stays | 90 days
  ICU stays
Hospital stays | 90 days
  Hospital stays
re-hospitalization rate | 90 days
  re-hospitalization rate
SOFA score | at days -1, 7, 14 and 28
  SOFA score
all-cause mortality | 90 days
  all-cause mortality
ICU mortality | 90 days
  ICU mortality
28-day ventilator-free days | 28-day
  28-day ventilator-free days
28-day ICU-free days | 28-day
  28-day ICU-free days
28-day CRRT-free days | 28-day
  28-day CRRT-free days
28-day Vasoactive agents-free days | 28-day
  28-day Vasoactive agents-free days
Septic shock | 28-day
  The incidence of septic shock
Sepsis heart injury | 28-day
  Ejection fraction<50% and left ventricular ejection fraction (LVEF) decreased by 10% from baseline，changes in biomarkers such as CKMB、cTNI caused by sepsis
Sepsis renal injury | 28-day
  Changes in biomarkers such as creatinine caused by sepsis
Sepsis liver injury | 28-day
  Changes in biomarkers such as ALT，AST caused by sepsis
Out-of-hospital mortality rate | Discharge for one year
  Mortality rate within one year after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Ji'nan, Shandong, China